CLINICAL TRIAL: NCT01822171
Title: Multi-Disciplinary Discharge Counseling and MTM Services After Discharge for Heart Failure Patients
Brief Title: Discharge Counseling and Medication Therapy Management (MTM) Services After Discharge for Heart Failure Patients
Acronym: MTM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll and study intended patient population.
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PSPH-002-Pharm
Record Dates: First submitted 2013-01-07; First posted 2013-04-02 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Medication Therapy Management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Discharge counseling and MTM follow-up (Experimental): At the time of hospital discharge the subject will receive:
  * Discharge medication counseling from a pharmacist
  * Home medication if needed
  * Approximately 7 days after hospital discharge the subject have a Follow-up visit at Medication Therapy Management clinic.
  Interventions: Other: Discharge medication counseling from a pharmacist; Other: Home medication if needed; Other: Follow-up visit at Medication Therapy Management clinic

INTERVENTIONS:
Other: Discharge medication counseling from a pharmacist — Patient will be educated about proper dosing instructions, potential side effects, and when to recontact the treating physician office.
Other: Home medication if needed — Patient will be provided with medication to take home, when needed.
Other: Follow-up visit at Medication Therapy Management clinic — This comprehensive Medication Therapy Management clinic follow-up visit is scheduled for 7 days post hospital discharge. The approximately 1 hour visit is scheduled with a pharmacist to review current drug therapy and make recommendations, if needed, to improve medication utilization.

SUMMARY:
Readmission to a hospital shortly after discharge is a common and costly problem. In the United States patients with a diagnosis of heart failure currently experience an elevated 30 day readmission rate of approximately 20%. By providing patients with medication related counseling at discharge by a pharmacist, home medications at discharge, and seeing the patient again in a pharmacist-run Medication Therapy Management (MTM) clinic 7 days after discharge, the study anticipates achieving its primary goal of showing a reduction in the readmission rate. Secondary goals are: 1) to determine patients understanding of the medication they are taking, 2) to evaluate satisfaction with the comprehensive discharge counseling service, and 3) determine the number of interventions made and benefit of the MTM clinic.

DETAILED DESCRIPTION:
The active arm of this study (medication related hospital discharge counseling by a pharmacist, home medications, and 7 day follow-up visit at a pharmacist run MTM clinic) is available to all subjects. To study the primary goal of reducing the 30 day readmission rate the data obtained from the active arm subjects will be compared to a match group of hospitalized patients that were previously discharged with a diagnosis of heart failure. The data for all secondary study goals will be obtained directly from the active arm subjects.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with high risk for readmission.
* Enroll in study prior to hospital discharge.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Reduction in hospital readmissions | 30 day
  The readmission rate for the 50 subjects involved in this study will be compared to an equal number patients retrospectively reviewed from a 2011 patient list and matched for heart failure severity. The primary outcome will based on a comparison of the ratio of patients readmitted to the hospital before the discharge instruction program started and after.

SECONDARY OUTCOMES:
Patient assessment of home medications knowledge at time of hospital discharge | 3 days
  Post hospital discharge the subject are asked to rate their knowledge regarding the medication they are taking at home on a scale of 1 to 10. The data obtained in this study will be compared to the same data and patient matched population obtained in 2011.
Patient satisfaction with comprehensive discharge counseling service. | 7 Days
  The satisfaction survey consists of five interview questions, where the subject subjectively scores each question on a scale of 1 to 10, developed specifically for this study.
Number of interventions made at the MTM clinic. | 7 Days.
  The number of drug related therapy interventions the pharmacist makes during the 7 day follow-up visit will be counted. Interventions may include: identifying: an inappropriate drug, inappropriate dose, duplication of medications, or a missing medication to optimize drug therapy.
Types of interventions made at the MTM clinic. | 7 days
  The types of intervention the pharmacist may work on during the 7 day follow-up visit include inappropriate drug, inappropriate dose, duplication of medications, missing medication to optimize drug therapy. Other types of interventions may be revealed during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hoekstra, Pharm.D., Principal Investigator — Providence St. Peter Hospital
Locations (2):
- United States (2):
  - Providence Centralia Hospital, Centralia, Washington
  - Providence St. Peter Hospital, Olympia, Washington